CLINICAL TRIAL: NCT04078412
Title: A Prospective Registry for Nontuberculous Mycobacterial Pulmonary Disease
Brief Title: A Registry for Nontuberculous Mycobacterial Pulmonary Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0958
Record Dates: First submitted 2019-08-29; First posted 2019-09-06 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Nontuberculous Mycobacterial Pulmonary Disease
Keywords: Nontuberculous mycobacteria; pulmonary; cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, urine, RNA and DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NTM pulmonary disease: Cohort Description: adults NTM pulmonary disease patients diagnose by criteria of American thoracic society guideline

SUMMARY:
Background:

NTM(Nontuberculous mycobacteria) pulmonary disease is increasing worldwidely, however the diagnosis and treatment of NTM pulmonary disease still has multiple obstacles. The initiation of treatment is not necessary for all patients with NTM pulmonary disease. In addition, the drugs for treatment of NTM pulmonary disease is not enough.

objective. The aim of this prospective registry for Nontuberculous mycobacterial pulmonary disease is to register the NTM pulmonary patients and analysis of the treatment outcome based on the species and to collect the blood and urine samples from the patients for exploring the biomarker for diagnosis and monitoring the NTM pulmonary disease and collect the nontuberculous mycobacterium.

Methods:

1. informed consents
2. register in cohort and collect the clinical information and serum, plasma, urine and mycobacteria
3. follow up 6 months to 1year based on the clinical situation

Analysis:

1. treatment outcome based on NTM-NET consensus statement
2. exploration of biomarker for progression and monitoring of treatment response

ELIGIBILITY:
Inclusion Criteria:

1. age 20 or more than 20 years
2. diagnosed by ATS criteria for NTM pulmonary disease

Exclusion Criteria:

1) not specific

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpaient clinic and hospitalzed patients in tertiary referral hospital
Sampling Method: Non-Probability Sample
Enrollment: 114 (Estimated)
Dates: Start 2017-11-21 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
treatment outcome based on NTM-NET consensus statement | At the end of the treatment or 12months after treatment
  1. For patients who need the treatment for NTM pulmonary disease : treatment outcome based on the NTM -NET consensus : microbiologic results, clinical symptoms and radiologic results
  2. For patients who don't need the treatment for NTM pulmonary disease : progression of NTM-PD defined by clinical, microbiotic and radiologic results.

SECONDARY OUTCOMES:
biomarker for disease progression: RNA sequence analysis | at the beginning of the treatment
  exploration for various biomarkers with RNA sequence analysis
biomarker for disease progression: metabolomic analysis | at the beginning of the treatment
  exploration for various biomarkers with metabolomic analysis
biomarker for disease progression: RNA sequence analysis | at the end of the treatment (through study completion, an average of 12 to 15month after treatment)
  exploration for various biomarkers with RNA sequence analysis
biomarker for disease progression: metabolomic analysis | at the end of the treatment (through study completion, an average of 12 to 15month after treatment)
  exploration for various biomarkers with metabolomic analysis
biomarker for monitoring of treatment response: RNA sequence analysis | at the beginning of the treatment
  exploration for various biomarkers with RNA sequence analysis
biomarker for monitoring of treatment response: metabolomic analysis | at the beginning of the treatment
  exploration for various biomarkers with metabolomic analysis
biomarker for monitoring of treatment response: RNA sequence analysis | at the end of the treatment (through study completion, an average of 12 to 15month after treatment)
  exploration for various biomarkers with RNA sequence analysis
biomarker for monitoring of treatment response: metabolomic analysis | at the end of the treatment (through study completion, an average of 12 to 15month after treatment)
  exploration for various biomarkers with metabolomic analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Yonsei University College of Medicine Division of Pulmonology, Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No